CLINICAL TRIAL: NCT07388524
Title: Evaluating Adjuvant Atezolizumab or Atezolizumab and Hyaluronidase-TQJS to Prevent Recurrence in Stage I Non-Small Cell Lung Cancer (NSCLC): A Randomized Phase III Trial (AASI-NSCLC)
Brief Title: Testing the Impact of an Anti-Cancer Drug, Atezolizumab, After Surgery to Prevent Early Stage Non-small Cell Lung Cancer From Returning, AASI-NSCLC Trial
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2026-00505; NCI-2026-00505 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A082302 (Other: Alliance for Clinical Trials in Oncology); A082302 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2026-02-04; First posted 2026-02-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Hyaluronoglucosaminidase; Specimen Handling; Watchful Waiting; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (observation) (Active Comparator): Patients undergo observation for 1 year. Patients also undergo CT and optional collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Patient Observation
- Arm B (atezolizumab) (Experimental): Patients receive atezolizumab IV over 60 minutes or atezolizumab and recombinant human hyaluronidase SC over 7 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for up to 1 year (17 cycles) in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and optional collection of blood samples throughout the trial.
  Interventions: Biological: Atezolizumab; Biological: Atezolizumab and Recombinant Human Hyaluronidase; Procedure: Biospecimen Collection; Procedure: Computed Tomography

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
  Arms: Arm B (atezolizumab)
Biological: Atezolizumab and Recombinant Human Hyaluronidase — Given SC
  Other Names: Atezolizumab + rHuPH20; Atezolizumab and Hyaluronidase; Atezolizumab and Hyaluronidase-tqjs; Atezolizumab and Recombinant Human Hyaluronidase-tqjs; Atezolizumab with rHuPH20; Atezolizumab-rHuPH20; atezolizumab/Hyaluronidase-tqjs; Atezolizumab/rHuPH20 Co-formulation; Recombinant Human Hyaluronidase Mixed with Atezolizumab; Tecentriq Hybreza; Tecentriq/rHuPH20
  Arms: Arm B (atezolizumab)
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Other: Patient Observation — Undergo observation
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
  Arms: Arm A (observation)

SUMMARY:
This phase III trial compares the effect of atezolizumab (or atezolizumab and recombinant human hyaluronidase) to standard observation for preventing cancer return after surgery (recurrence) in patients who have undergone a complete surgical removal (resection) of stage I non-small cell lung cancer (NSCLC). Patients who have undergone resection for lung cancer are typically followed by observation or active surveillance, which involves closely watching a patient's condition but not giving treatment unless there are changes in test results. During active surveillance, patients are given certain exams and tests done on a regular schedule. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Atezolizumab and recombinant human hyaluronidase is a formulation of atezolizumab combined with an enzyme called hyaluronidase, which helps increase tissue absorption of the drug. Giving atezolizumab or atezolizumab and recombinant human hyaluronidase after resection may be effective for preventing NSCLC recurrence, and may be a better approach to treating patients with stage I NSCLC than the usual observation approach.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare disease-free survival (DFS) in the intent-to-treat patient population, among patients randomized to receive atezolizumab for one year (Arm B) versus (vs.) observation (Arm A).

SECONDARY OBJECTIVES:

I. To compare overall survival (OS) between patients randomized to atezolizumab versus observation.

II. To compare recurrence-free survival (RFS) between patients randomized to atezolizumab versus observation.

III. To compare lung-cancer-specific OS between patients randomized to atezolizumab versus observation.

IV. To compare rates of loco-regional recurrences between patients randomized to atezolizumab versus observation.

V. To compare rates of distant recurrences between patients randomized to atezolizumab versus observation.

VI. To compare adverse event rates (AEs) via Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5 between patients randomized to atezolizumab versus observation.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients undergo observation for 1 year. Patients also undergo computed tomography (CT) and optional collection of blood samples throughout the trial.

ARM B: Patients receive atezolizumab intravenously (IV) over 60 minutes or atezolizumab and recombinant human hyaluronidase subcutaneously (SC) over 7 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for up to 1 year (17 cycles) in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and optional collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up at 30 days (patients in Arm B only), then every 6 months for 3 years and then annually thereafter for an additional 7 years (10 years total).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically stage IA3 or IB NSCLC per American Joint Committee on Cancer (AJCC) Cancer Staging Manual, 9th edition

  * Note: Tumors with any histology are allowed including both squamous and non-squamous subtypes, except those containing small-cell morphology. Non-squamous histology includes adenocarcinoma, large cell neuroendocrine, poorly differentiated tumors and adenosquamous, etc
* Patient must have undergone complete surgical resection with negative margins (complete R0 resection). Surgical resection must be lobectomy or higher, unless the tumor measured no more than 2 cm based on clinical staging, where sub-lobar resection, e.g., wedge or segmentectomy, will be acceptable

  * Note: For patients who underwent sub-lobar resection for clinical tumors size of ≤ 2.0 cm, must have CT chest confirming tumor size within 60 days of surgical resection. Patients who received a lobectomy or higher do not require to fulfill this imaging criteria
* Patient must have undergone adequate nodal sampling as defined by Commission on Cancer, 2020 Standard. Adequate nodal sampling includes pathological evaluation of at least one (named and/or numbered) hilar station (level 10 or higher) and at least three distinct (named and or numbered) mediastinal stations (level 2-9)
* PD-L1 immunohistochemistry showing tumor proportion score (TPS) ≥ 50%, by an Food and Drug Administration (FDA)-approved assay including but not limited to SP263, SP142, 22C3, 28-8, performed either on surgical specimen or biopsy specimen
* No EGFR exon 19 deletion (del) or L858R mutation or ALK fusion; molecular testing may have been performed either on surgical specimen or biopsy specimen. Tumors with purely squamous histology are not required to undergo EGFR or ALK gene testing
* Patient to be registered to A082302 no earlier than 21 days and no later than 77 days from surgical resection
* Recovered from surgical resection as determined by the treating provider or the investigator
* No prior neoadjuvant or adjuvant therapy for current lung cancer diagnosis
* Patient must NOT have uncontrolled intercurrent illness, including but not limited to serious ongoing or active infection, symptomatic congestive heart failure (New York Heart Association [NYHA] class ≥ III), unstable angina, or unstable arrhythmia
* No current pneumonitis or history of (non-infectious) pneumonitis that required steroids or history of interstitial lung disease (ILD)
* No active auto-immune disease that has required systemic treatment within the last 2 years (e.g., disease modifying agents, corticosteroids, or immunomodulatory agents). Replacement therapy (e.g., thyroid for history of autoimmune thyroiditis, insulin for type I or II diabetes, corticosteroids for adrenal or pituitary insufficiency) is not considered a form of systemic treatment
* No known hypersensitivity (≥ grade 3) to atezolizumab and/or any of its excipients
* No live vaccine within 30 days prior to registration. Examples include but are not limited to: measles, mumps, rubella, varicella, yellow fever, Bacillus Calmette-Guerin (BCG), typhoid, nasally administered influenza
* No history of prior allogeneic bone marrow, stem cell, or solid organ transplant
* Patient has not received continuous systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalents) or other immunosuppressive medications within 14 days prior to registration, with the following exceptions:

  * Inhaled or topical steroids and adrenal replacement doses ≤ 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, if < 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen or chronic obstructive pulmonary disease [COPD] exacerbation) is permitted
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (or Karnofsky ≥ 60%)
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN), except patients with Gilbert syndrome who can have total bilirubin < 3.0 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 3 x upper limit of normal (ULN)
* Creatinine clearance ≥ 30 mL/min (using standard Cockcroft-Gault formula, unless measured creatinine clearance [CrCl] is available and meet the specified threshold)
* Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects

  * Therefore, for women of childbearing potential only, a negative urine or serum pregnancy test done ≤ 7 days prior to registration is required
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial

  * HIV: Patients with known HIV infection on effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration are eligible for this trial. Patients with no known history of HIV do not require any testing
* Hepatitis B and hepatitis C: No active hepatitis B (defined as negative for hepatitis B [HepB] deoxyribonucleic acid [DNA], and positive for HepB surface antibody) or hepatitis C (defined as hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] detected) infection. If there is a history of either infection, patient should be negative for active disease, for hepatitis B negative for hepatitis B virus surface antigen (HBsAg), and for hepatitis C - negative for HCV RNA (qualitative). Patients with no known history of chronic hepatitis do not require any testing
* No active infection requiring systemic therapy
* Cardiac function: Patients with known history or current symptoms of heart failure, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification. To be eligible for this trial, patients should be class 2B or better

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2026-04-09 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | From randomization to disease recurrence, second lung primary, or death, assessed up to 10 years
  Distributions of survival time between treatment arms will be compared with a one-sided stratified log-rank test. The rates at various timepoints and medians for each arm will be estimated using the Kaplan-Meier estimator. The 95% confidence interval will be calculated using Greenwood's formula and based on a log-log transformation applied to the survival function. Hazard ratios will be estimated using a stratified Cox regression model. Multivariable Cox models will be used to evaluate the treatment effect on survival time and its interaction with baseline covariates, including stage, systemic regimen, histology, and performance status.

SECONDARY OUTCOMES:
Overall survival | From randomization to death, assessed up to 10 years
  Distributions of survival time between treatment arms will be compared with a one-sided stratified log-rank test.
Lung cancer-specific survival | Up to 10 years
  Distributions of survival time between treatment arms will be compared with a one-sided stratified log-rank test.
Recurrence-free survival | From randomization to recurrence or death, assessed up to 10 years
  Recurrence will be characterized as loco-regional or distant. Distributions of survival time between treatment arms will be compared with a one-sided stratified log-rank test.
Rate of loco-regional recurrence | Up to 10 years
  Rates between arms will be compared with Fisher's exact test. The difference in recurrence rates between arms will be estimated by the Miettinen-Nurminen method, and its 95% confidence interval will be provided. Multivariable logistic regression will be used to evaluate the treatment effect on the recurrence rates while adjusting for significant baseline covariates.
Rate of distant recurrence | Up to 10 years
  Rates between arms will be compared with Fisher's exact test. The difference in recurrence rates between arms will be estimated by the Miettinen-Nurminen method, and its 95% confidence interval will be provided. Multivariable logistic regression will be used to evaluate the treatment effect on the recurrence rates while adjusting for significant baseline covariates.
Incidence of grade ≥ 3 adverse events | Up to 10 years
  The maximum grade for each type of adverse event will be summarized using Common Terminology Criteria for Adverse Events version 5. The frequency and percentage of grade ≥ 3 adverse events will be compared between the study arms using Fisher's exact test.

OTHER OUTCOMES:
Disease free survival by sex | Up to 10 years
  Estimates of disease-free survival and the corresponding 95% confidence intervals by sex will be provided.
Disease free survival by race | Up to 10 years
  Estimates of disease-free survival and the corresponding 95% confidence intervals by race will be provided.
Disease free survival by ethnicity | Up to 10 years
  Estimates of disease-free survival and the corresponding 95% confidence intervals by ethnicity will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Furqan, Principal Investigator — Alliance for Clinical Trials in Oncology

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm